CLINICAL TRIAL: NCT01116856
Title: Nutrition and Physical Activity Programs for Obesity Treatment (PRONAF)
Brief Title: Nutrition and Physical Activity for Obesity
Acronym: PRONAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Universidad Complutense de Madrid (Other); Hospital Universitario La Paz (Other); Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Pedro JoseBenito Peinado, PhD, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRONAF
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Overweight
Keywords: Exercise; Training; Obesity; Overweight; Body composition; Lipidic profile; Nutrition; Polymorphisms
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two phases, the first for overweight, and the second for obese people
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nutrition (Experimental): This groups will follow a diet.
  Interventions: Other: Exercise
- Nutrition + resistance training (Experimental): In this group, nutrition and resistance training will be combined.
  Interventions: Other: Exercise
- Nutrition + aerobic training (Experimental): In this group nutrition and aerobic training will be combined.
  Interventions: Other: Exercise
- Nutrition + mixed training (Experimental): In this group the nutrition will be combined with 50% of resistance training plus 50% of aerobic training.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Different groups will carry out different exercise protocols during 16 weeks under the same nutritional intervention.

SUMMARY:
At the present time, scientific consensus exists on obesity multifactorial etiopatogenia. As well, professionals and researchers agree that the treatment must approach several scopes, such as dietetic, physical activity, pharmacologic and surgical. These two last ones should not be the first election and must be reserved for those cases of morbid obesities or in case the previous ones have failed. The combination of diet and exercise is still not sufficiently studied, in special, the addition of strength training, as we propose in this project, for which established intervention protocols do not exist, and that could suppose an additional benefit in the reduction of risk factors.

Therefore, the objectives that we aim in this project are enumerated below:

* To discover which are the most effective training protocols and to determine what type of exercise combined with nutrition is more appropriate for obesity intervention programs.
* To establish the relationship between markers related with cardiovascular risk (adopokines and lipid profile) and the different intervention protocols proposed.
* To describe the influence of nine genetic polymorphisms (selected by their relationship with the energy expense and the physical yield) on the effect of different training protocols.
* To determine how important is body composition (fat mass and muscle mass mainly) in total daily energy expenditure.
* To establish rules of nutritional and exercise intervention that can be applied in public and private training centers. If the proposed objectives are fulfilled, this would contribute to an improvement in patients health in long term, along with an enormous saving in public health. Therefore, the purpose of this project is to propose new lines of intervention in overweight and obese adults that, until now, little have been investigated. This way, resistance training is proposed in combination with cardiovascular training and endocrinologic treatment. It fits to emphasize that, as far as we know, it is the first project of these characteristics, that puts in touch the public and private sector (hospitals, universities and fitness area), to establish standardized relations protocols to allow a close pursuit of obese patients.

ELIGIBILITY:
For Overweight phase:

Inclusion Criteria:

* Volunteers: men and women from Comunidad de Madrid (Zone 5 of Health System) who sign the informed consent.
* Ages 18 - 50 years old.
* Pre-menopausal.
* Body mass index (BMI) of 25 - 30 kg•m-2 (both included).
* Able to attend exercise classes 3 times per week (Monday, Wednesday and Friday). No plans for excessive travel. No plans to move from area for study period (January 2010 - June 2010, both included).
* Able to follow the nutritional treatment (avoid medication or substances known to interfere with body weight regulation, including anti-depressive medication, diuretics, etc., 15 days before study starts).
* Willing to not participate in other formal or informal weight loss program during the period of the study.
* Sedentary (less than once a week of training or two hours of physical activity class).

Exclusion Criteria:

* Smoking within six months, or use of tobacco or nicotine product.
* Women with irregular menstrual cycle (except with hormone therapy).
* Following a weight loss diet, vegetarians or food restriction due to religion.
* Self-reported weight loss or gain >5% in past 6 months.
* Are not pregnant, or haven´t been in the past six months. Are not currently nursing or planning to become pregnant during the study period (year 2010).
* Need a special diet by associated disease (celiac disease or chronic renal insufficiency).
* Have metabolic syndrome or fulfill three or more of the following criteria: abdominal obesity (waist diameter > 102 cm in men and > 88 cm in women), blood pressure ≥ 130/85 mm Hg, basal glycemia ≥ 110 mg/dL, triglyceride level > 150 mg/dL and C-HDL < 40 mg/dL in women and < 50 mg/dL in men.
* Diabetes.
* Anemia (Hct < 37%).
* Uncontrolled high blood pressure (Systolic > 160 mm Hg or diastolic > 100 mm Hg in rest). Current use of more than one anti-hypertensive medication.
* Substance abuse (drugs, alcohol…). High or moderate consumes of alcohol. More than 2 glasses to the day of any alcoholic substance. Current use of diuretics, beta blockers, steroids or blood thinners.
* Contraindication to exercise. Alterations, syndromes or diseases detected by electrocardiogram (EKG) o echocardiography. Have injuries o pathologies of the locomotive apparatus that prevent the correct execution of the exercises of the program. Any illness that would prevent participation in a moderate-intense exercise program.
* Have had cancer in the past 5 years, except skin cancer.
* Coronary artery disease, liver disease, pulmonary disease, renal disease or other systemic disorders.
* History or evidence of cardiovascular disease, alterations, syndromes or other mayor chronic illness. Have history of heart disease, heart attacks or heart surgery.
* Have any illness known to interfere with body weight loss: clinical depression, eating disorder (anorexia, bulimia, etc.), psychological diseases (schizophrenia, etc.), dementia or cognitive function decreased, hypothyroidism no controlled or history of genetic or chromosomal disorder.
* Have had bariatric surgery or stomach bypass surgery.
* Gross physical impairment.
* Blindness or retinopathy.

For Obese phase:

Inclusion Criteria:

* Volunteers: men and women from Comunidad de Madrid (Zone 5 of Health System) who sign the informed consent.
* Ages 18 - 50 years old.
* Pre-menopausal.
* Body mass index (BMI) of 30 - 35 kg•m-2 (both included).
* Able to attend exercise classes 3 times per week (Monday, Wednesday and Friday). No plans for excessive travel. No plans to move from area for study period (January 2011 - June 2011, both included).
* Able to follow the nutritional treatment (avoid medication or substances known to interfere with body weight regulation, including anti-depressive medication, diuretics, etc., 15 days before study starts).
* Willing to not participate in other formal or informal weight loss program during the period of the study.
* Sedentary (less than once a week of training or two hours of physical activity class).

Exclusion Criteria:

* Smoking within six months, or use of tobacco or nicotine product.
* Women with irregular menstrual cycle (except with hormone therapy).
* Following a weight loss diet, vegetarians or food restriction due to religion.
* Self-reported weight loss or gain >5% in past 6 months.
* Are not pregnant, or haven´t been in the past six months. Are not currently nursing or planning to become pregnant during the study period (year 2011).
* Need a special diet by associated disease (celiac disease or chronic renal insufficiency).
* Have metabolic syndrome or fulfill three or more of the following criteria: abdominal obesity (waist diameter > 102 cm in men and > 88 cm in women), blood pressure ≥ 130/85 mm Hg, basal glycemia ≥ 110 mg/dL, triglyceride level > 150 mg/dL and C-HDL < 40 mg/dL in women and < 50 mg/dL in men.
* Diabetes.
* Anemia (Hct < 37%).
* Uncontrolled high blood pressure (Systolic > 160 mm Hg or diastolic > 100 mm Hg in rest). Current use of more than one anti-hypertensive medication.
* Substance abuse (drugs, alcohol…). High or moderate consumes of alcohol. More than 2 glasses to the day of any alcoholic substance. Current use of diuretics, beta blockers, steroids or blood thinners.
* Contraindication to exercise. Alterations, syndromes or diseases detected by electrocardiogram (EKG) o echocardiography. Have injuries o pathologies of the locomotive apparatus that prevent the correct execution of the exercises of the program. Any illness that would prevent participation in a moderate-intense exercise program.
* Have had cancer in the past 5 years, except skin cancer.
* Coronary artery disease, liver disease, pulmonary disease, renal disease or other systemic disorders.
* History or evidence of cardiovascular disease, alterations, syndromes or other mayor chronic illness. Have history of heart disease, heart attacks or heart surgery.
* Have any illness known to interfere with body weight loss: clinical depression, eating disorder (anorexia, bulimia, etc.), psychological diseases (schizophrenia, etc.), dementia or cognitive function decreased, hypothyroidism no controlled or history of genetic or chromosomal disorder.
* Have had bariatric surgery or stomach bypass surgery.
* Gross physical impairment.
* Blindness or retinopathy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Body composition | After 16 weeks of intervention
Health status | After 16 weeks of intervention
Cardiorespiratory fitness | After 16 weeks of intervention

SECONDARY OUTCOMES:
Quality of life | After 16 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Benito, PhD, Principal Investigator — Department of Health and Human Performance, Universidad Politécnica de Madrid
Locations (2):
- Spain (2):
  - Pedro J. Benito Peinado, Madrid
  - Facultad de Ciencias de la Actividad Física y del Deporte, Madrid

REFERENCES:
- [Derived] Cupeiro R, Benito P, Amigo T, Gonzalez-Lamuno D. The association of SLC16A1 (MCT1) gene polymorphism with body composition changes during weight loss interventions: A randomized trial with sex-dependent analysis. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-12. doi: 10.1139/apnm-2024-0246. PMID 39787575
- [Derived] Benito PJ, Lopez-Plaza B, Bermejo LM, Peinado AB, Cupeiro R, Butragueno J, Rojo-Tirado MA, Gonzalez-Lamuno D, Gomez-Candela C, On Behalf Of The Pronaf Study Group. Strength plus Endurance Training and Individualized Diet Reduce Fat Mass in Overweight Subjects: A Randomized Clinical Trial. Int J Environ Res Public Health. 2020 Apr 10;17(7):2596. doi: 10.3390/ijerph17072596. PMID 32290136
- [Derived] Benito PJ, Cupeiro R, Peinado AB, Rojo MA, Maffulli N; PRONAF Study Group. Influence of previous body mass index and sex on regional fat changes in a weight loss intervention. Phys Sportsmed. 2017 Nov;45(4):450-457. doi: 10.1080/00913847.2017.1380500. Epub 2017 Oct 5. PMID 28914104
- [Derived] Castro EA, Judice PB, Silva AM, Teixeira PJ, Benito PJ. Sedentary behavior and compensatory mechanisms in response to different doses of exercise-a randomized controlled trial in overweight and obese adults. Eur J Clin Nutr. 2017 Dec;71(12):1393-1398. doi: 10.1038/ejcn.2017.84. Epub 2017 May 31. PMID 28561039
- [Derived] Benito PJ, Alvarez-Sanchez M, Diaz V, Morencos E, Peinado AB, Cupeiro R, Maffulli N; PRONAF Study Group. Cardiovascular Fitness and Energy Expenditure Response during a Combined Aerobic and Circuit Weight Training Protocol. PLoS One. 2016 Nov 10;11(11):e0164349. doi: 10.1371/journal.pone.0164349. eCollection 2016. PMID 27832062
- [Derived] Benito PJ, Bermejo LM, Peinado AB, Lopez-Plaza B, Cupeiro R, Szendrei B, Calderon FJ, Castro EA, Gomez-Candela C; PRONAF Study Group. Change in weight and body composition in obese subjects following a hypocaloric diet plus different training programs or physical activity recommendations. J Appl Physiol (1985). 2015 Apr 15;118(8):1006-13. doi: 10.1152/japplphysiol.00928.2014. Epub 2015 Feb 26. PMID 25722378
- [Derived] Rojo-Tirado MA, Benito PJ, Atienza D, Rincon E, Calderon FJ. Effects of age, sex, and treatment on weight-loss dynamics in overweight people. Appl Physiol Nutr Metab. 2013 Sep;38(9):967-76. doi: 10.1139/apnm-2012-0441. Epub 2013 Apr 30. PMID 23905663
- [Derived] Morencos E, Romero B, Peinado AB, Gonzalez-Gross M, Fernandez C, Gomez-Candela C, Benito PJ; PRONAF study group. Effects of dietary restriction combined with different exercise programs or physical activity recommendations on blood lipids in overweight adults. Nutr Hosp. 2012 Nov-Dec;27(6):1916-27. doi: 10.3305/nh.2012.27.6.6057. PMID 23588439
- [Derived] Zapico AG, Benito PJ, Gonzalez-Gross M, Peinado AB, Morencos E, Romero B, Rojo-Tirado MA, Cupeiro R, Szendrei B, Butragueno J, Bermejo M, Alvarez-Sanchez M, Garcia-Fuentes M, Gomez-Candela C, Bermejo LM, Fernandez-Fernandez C, Calderon FJ. Nutrition and physical activity programs for obesity treatment (PRONAF study): methodological approach of the project. BMC Public Health. 2012 Dec 21;12:1100. doi: 10.1186/1471-2458-12-1100. PMID 23259716
- [Derived] Loria-Kohen V, Fernandez-Fernandez C, Bermejo LM, Morencos E, Romero-Moraleda B, Gomez-Candela C. Effect of different exercise modalities plus a hypocaloric diet on inflammation markers in overweight patients: a randomised trial. Clin Nutr. 2013 Aug;32(4):511-8. doi: 10.1016/j.clnu.2012.10.015. Epub 2012 Nov 6. PMID 23177481